CLINICAL TRIAL: NCT02920749
Title: Recovery Profiles and Costs in Sevoflurane and Propofol Based Anaesthesia
Brief Title: Study of Anaesthesia Costs and Recovery Profiles
Acronym: SACRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Timea Bocskai, Assistant Professor, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 316-2336/KK15
Record Dates: First submitted 2016-09-25; First posted 2016-09-30 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Anaesthesia
Keywords: anaesthesia; costs; recovery profiles

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sevoflurane group A (Other): Anaesthesia was maintained with sevoflurane (1-2% end-tidal concentration, MAC 1.0-1.5) in 50% air and 50% oxygen mixture.
  Interventions: Drug: Sevoflurane group A
- Sevoflurane group B (Other): Anaesthesia was maintained with sevoflurane (1-2% end-tidal concentration, MAC 1.0-1.5) in 50% air and 50% oxygen mixture. Sevoflurane dosing was set to maintain target BIS levels of 40 to 60 and MAP for controlled hypotension within 60-85 mmHg.
  Interventions: Drug: Sevoflurane group B
- Propofol group C (Other): During anaesthesia TIVA was applied with a protocol (6 to 8 mg/kg/h propofol).
  Interventions: Drug: Propofol group C
- Propofol group D (Other): Propofol dosing was set to maintain target BIS levels of 40 to 60 and MAP for controlled hypotension within 60-85 mmHg.
  Interventions: Drug: Propofol group D

INTERVENTIONS:
Drug: Sevoflurane group A — In this group anaesthesia was maintained with sevoflurane. Initial and maintenance fresh gas flow was 4 and 1 l/min, respectively. Sevoflurane dosing was adjusted for the same MAP range.
  Other Names: Sevorane anaesthesia
  Arms: Sevoflurane group A
Drug: Sevoflurane group B — In this group anaesthesia was maintained with sevoflurane. Initial and maintenance fresh gas flow was 4 and 1 l/min, respectively. Sevoflurane dosing was set to maintain target BIS levels of 40 to 60 and MAP for controlled hypotension within 60-85 mmHg.
  Other Names: Sevorane anaesthesia with BIS and TOF monitoring
  Arms: Sevoflurane group B
Drug: Propofol group C — In this group anaesthesia was maintained with propofol. Propofol was administered according to protocol. Propofol dosing was adjusted for the same MAP range.
  Other Names: Propofol anaesthesia
  Arms: Propofol group C
Drug: Propofol group D — In this group anaesthesia was maintained with propofol. Propofol dosing was set to maintain target BIS levels of 40 to 60 and MAP for controlled hypotension within 60-85 mmHg.
  Other Names: Propofol anaesthesia with BIS and TOF monitoring
  Arms: Propofol group D

SUMMARY:
The purpose of this study is to compare the perioperative hemodynamic parameters, recovery profiles and cost containment of sevoflurane and propofol based general anesthesia for otorhinolaryngeal surgery.

DETAILED DESCRIPTION:
Sevoflurane and propofol are two basic drugs in the maintenance of anaesthesia. In this study we compared the perioperative hemodynamic parameters, recovery profiles and cost containment of sevoflurane and propofol based general anaesthesia for otorhinolaryngeal surgery. Patients were equally divided into four anaesthetic subgroups. In groups A and C anaesthesia was based on sevoflurane or propofol, respectively, without bispectral index (BIS) and train-of-for monitor (TOF) monitoring. In groups B and D anaesthesia was based on sevoflurane or propofol, respectively, with BIS and TOF monitoring. Drug consumption, recovery profiles and anaesthesia costs were analysed.

ECG, main arterial pressure (MAP), heart rate, oxygen saturation of peripheral haemoglobin (SpO2), pressure of end-tidal carbon dioxide was monitored continuously and registered at 5 min intervals during anaesthesia. Each group received propofol for anaesthesia induction. In group A and B anaesthesia was maintained with sevoflurane, in groups C and D with propofol. In groups B and D the depth of anaesthesia (BIS® Quatro Brain Monitoring Sensor, Covidien) and the neuromuscular blocking status (Infinity®, Trident® NMT SmartPod®, Dräger Medical) were monitored too. BIS and TOF values were recorded at 5 min intervals.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status grade I or II who were scheduled for elective otorhinolaryngological surgery.

Exclusion Criteria:

* Individuals with a history of bronchial asthma, chronic obstructive pulmonary disease, epilepsy, psychiatric illness, cerebrovascular or congenital neuromuscular disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Csaba Loibl, MD, Study Chair — Department of Anesthesiology and Intensive Therapy, University of Pecs, Hungary; Zoltan Vamos, MD, PhD, Study Chair — Department of Anesthesiology and Intensive Therapy, University of Pecs, Hungary; Gabor Woth, MD, PhD, Study Chair — Department of Anesthesiology and Intensive Therapy, University of Pecs, Hungary; Lajos Bogar, MD, PhD, DSc, Study Director — Department of Anesthesiology and Intensive Therapy, University of Pecs, Hungary; Laszlo Lujber, MD, PhD, Study Director — Department of Otorhinolaryngology, University of Pecs, Hungary
Locations (1):
- Tímea Bocskai, Pécs, Ifjusag Street 13., Hungary

IPD SHARING:
Plan to Share IPD: Yes
Data of primary outcome measures will be made available within one month of study completion

REFERENCES:
- [Derived] Bocskai T, Loibl C, Vamos Z, Woth G, Molnar T, Bogar L, Lujber L. Cost-effectiveness of anesthesia maintained with sevoflurane or propofol with and without additional monitoring: a prospective, randomized controlled trial. BMC Anesthesiol. 2018 Jul 28;18(1):100. doi: 10.1186/s12871-018-0563-z. PMID 30055562

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study we compared the perioperative hemodynamic parameters, recovery profiles and cost containment of sevoflurane and propofol based general anaesthesia with controlled hypotension for otorhinolaryngeal surgery.
Pre-assignment Details: We studied patients with ASA physical status I or II, their age between was between 18 and 65 years. Individuals with a history of pulmonary, psychiatric, cerebrovascular or congenital neuromuscular disease were excluded from the study. Patients were blocked randomised to one of four anaesthetic treatment groups with closed envelops.
Groups:
- Group A: Anaesthesia was maintained with sevoflurane. Initial and maintenance fresh gas flow was 4 and 1 l/min, respectively. Sevoflurane and fentanyl dosing was adjusted for the same MAP range for controlled hypotension within 60-85 mmHg. Atracurium was administered at regular intervals.
- Group B: In this group anaesthesia was maintained with sevoflurane. Initial and maintenance fresh gas flow was 4 and 1 l/min, respectively. The depth of anaesthesia (BIS® Quatro Brain Monitoring Sensor, Covidien) and the neuromuscular blocking status (Infinity®, Trident® NMT SmartPod®, Dräger Medical) was monitored too. Sevoflurane and fentanyl dosing was set to maintain target BIS levels of 40 to 60 and MAP for controlled hypotension within 60-85 mmHg. Neuromuscular blocking was maintained with a TOF monitor at the level of one or no response.
- Group C: Anaesthesia was maintained with propofol. Propofol was administered according to protocol. Propofol and fentanyl dosing was adjusted for the same MAP range. Atracurium was administered at regular intervals.
- Group D: In this group anaesthesia was maintained with propofol. The depth of anaesthesia (BIS® Quatro Brain Monitoring Sensor, Covidien) and the neuromuscular blocking status (Infinity®, Trident® NMT SmartPod®, Dräger Medical) was monitored too. Propofol and fentanyl dosing was set to maintain target BIS levels of 40 to 60 and MAP for controlled hypotension within 60-85 mmHg. Neuromuscular blocking was maintained with a TOF monitor at the level of one or no response.
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D
Started | 30 | 30 | 30 | 30
Completed | 30 | 30 | 30 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: General anaesthesia was maintained with sevoflurane.
- Group B: Anaesthesia was maintained with sevoflurane and the depth of anaesthesia (BIS® Quatro Brain Monitoring Sensor, Covidien) and the neuromuscular blocking status (Infinity®, Trident® NMT SmartPod®, Dräger Medical) was monitored too.
- Group C: General anaesthesia was maintained with propofol.
- Group D: Anaesthesia was maintained with propofol and the depth of anaesthesia (BIS® Quatro Brain Monitoring Sensor, Covidien) and the neuromuscular blocking status (Infinity®, Trident® NMT SmartPod®, Dräger Medical) was monitored too.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 30 | 30 | 120
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 19 | 16 | 65
  Male | 16 | 14 | 11 | 14 | 55
Region of Enrollment [Number; unit: participants]
  Hungary | 30 | 30 | 30 | 30 | 120

OUTCOME MEASURES:

1. Primary Outcome: Drug Consumption
Description: drugs of sevoflurane or total intravenous anaesthesia without or with BIS and TOF monitoring : fentanyl, sevoflurane, propofol 1%, atracurium in milligrams
Time Frame: at induction one dose and during anaesthesia mg/1 hour
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Group A: Fentanyl consumption was studied during sevoflurane anaesthesia. It was registered in milligram.
- Group B: Fentanyl consumption was studied during sevoflurane anaesthesia with BIS and TOF monitoring. It was registered in milligram.
  .
- Group C: Fentanyl consumption was studied during total intravenous anaesthesia. It was registered in milligram.
- Group D: Fentanyl consumption was studied during total intravenous anaesthesia with BIS and TOF monitoring. It was registered in milligram.
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 30 | 30 | 30 | 30
mg
  fentanyl at induction | 0.0983 (0.0091) | 0.1033 (0.0183) | 0.0991 (0.0046) | 0.0992 (0.0103)
  propofol at induction | 196.3 (46.9) | 166.4 (35.2) | 194.3 (18.9) | 147.3 (30.2)
  atracurium at induction | 38.3 (4.2) | 37.3 (6.7) | 36.0 (5.7) | 37.7 (7.0)
  fentanyl during anaesthesia | 0.0546 (0.0269) | 0.0598 (0.0389) | 0.0898 (0,0428) | 0.0947 (0.0340)
  sevoflurane during anesthesia | 11400 (2800) | 14800 (12400) | 0 (0) | 0 (0)
  propofol during anesthesia | 0 (0) | 0 (0) | 1185.5 (320.9) | 1082.1 (297.9)
  atracurium during anaesthesia | 8.3 (3.7) | 7.4 (4.7) | 8.5 (4.7) | 8.9 (6.1)
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C vs Group D; Statistical analysis was carried out with SPSS version 21 for Windows (IBM Corporation) software. All data are expressed as means ± SD. Mann-Whitney test was performed to assess the differences between patient subgroups; Test type: Superiority or Other; p < 0.05, ANOVA — The P value less than 0.05 was considered to be significant. With type I α = 5% and with type II (power) of 90%, we therefore needed 27 patients/group

2. Secondary Outcome: Costs of Anaesthesia
Description: total cost of drugs (midazolam, propofol 1%, sevoflurane, atracurium, diclofenac, nalbuphin and antidotes) and disposable cost in euros
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: euros
Units Other Than Participants: total cost of anaesthesia
Groups:
- Group A: Drugs at induction were: fentanyl, propofol 1%, atracurium. Anaesthesia was maintained with sevoflurane, fentanyl and atracurium.
  Cost was calculated in euros/1 hour. Disposable cost was calculated in euros.
- Group B: Drugs at induction were: fentanyl, propofol 1%, atracurium. Anaesthesia was maintained with sevoflurane, fentanyl and atracurium.
  Cost was calculated in euros/1 hour. Disposable cost was calculated in euros. In this group BIS sensor and TOF monitoring was used.
- Group C: Drugs at induction were: fentanyl, propofol 1%, atracurium. Anaesthesia was maintained with propofol 1%, fentanyl and atracurium.
  Cost was calculated in euros/1 hour. Disposable cost was calculated in euros.
- Group D: Drugs at induction were: fentanyl, propofol 1%, atracurium. Anaesthesia was maintained with propofol, fentanyl and atracurium.
  Cost was calculated in euros/1 hour. Disposable cost was calculated in euros. In this group BIS sensor and TOF monitoring was used.
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 30 | 30 | 30 | 30
Number analyzed (total cost of anaesthesia) | 30 | 30 | 30 | 30
euros
  total drug cost | 8.84 (4.11) | 7.86 (3.54) | 8.33 (3.02) | 7.52 (2.49)
  total disposable cost | 6.49 (0.11) | 23.25 (0.12) | 8.09 (0.07) | 24.76 (0.19)
  total cost of anaesthesia | 12.15 (5.32) | 19.95 (8.53) | 13.23 (4.23) | 22.11 (8.08)
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C vs Group D; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Group A: Anaesthesia was maintained with sevoflurane (1-2% end-tidal concentration, MAC 1.0-1.5) in 50% air and 50% oxygen mixture.
  Fentanyl consumption was studied during anaesthesia. It was registered in milligram.
- Group B: Anaesthesia was maintained with sevoflurane (1-2% end-tidal concentration, MAC 1.0-1.5) in 50% air and 50% oxygen mixture.
  Fentanyl consumption was studied during anaesthesia. It was registered in milligram.
  .
- Group C; Group D: During anaesthesia TIVA was applied with a protocol (6 to 8 mg/kg/h propofol). Fentanyl consumption was studied during anaesthesia. It was registered in milligram.
Arm/Group | Group A | Group B | Group C | Group D
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 14/30 | 15/30 | 4/30 | 8/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=30) | Group B (N=30) | Group C (N=30) | Group D (N=30)
vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 1
other minor complications of anaesthesia (Cardiac disorders) | 13 | 13 | 3 | 7

LIMITATIONS AND CAVEATS:
This study is restricted to anaesthesia of otorhinolaryngological surgery with controlled hypotension. Therefore, we cannot draw any conclusions related to other surgeries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No